CLINICAL TRIAL: NCT03458663
Title: Single-blinded, Randomized Study Comparing Healing After Bascom's Cleft Lift Operation for Pilonidal Disease With or Without Prevena ™ and ACTIV.A.C ™ Therapy System
Brief Title: Randomized Trial Comparing Prevena and ActiV.A.C. System to Convetional Care After Bascom's Cleft Lift Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interrim analysis showed no effect or a tendency towards poorer out come in the Prevena group
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCTBCL2018
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized controlled trial .
Who Masked: Outcomes Assessor
Masking Description: Patients will be seen and the primary outcome assesed by a nurse in the out patient department who is blinded to the postoperative care the patient has recieved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevena (Experimental): Patients randomized to application of Prevena ™ and ACTIV.A.C ™ Therapy System 4-7 days post-operatively. Patients will return to the surgical day clinic to have the system removed either at day 7 or when/ if function ceases. Patients receive 3 days oral antibiotics postoperatively (Ciproxin 250 mg x 2 and Metronidazole 500 mg x 3). Sutures are removed at clinical control after 14 days and patients are seen again by BCL surgeon after 3 months and are discharged when completely healeddrainage and conventional wound dressing
  Interventions: Device: Prevena™ og ACTIV.A.C™ Therapy System.
- Conentional postoperative care (No Intervention): patients randomized to convetional postoperative regime with a penrose drain (passive) and a dry draping for 24 hours and after usage of sanitary pads. Patients receive 3 days oral antibiotics postoperatively (Ciproxin 250 mg x 2 and Metronidazole 500 mg x 3). Drain is removed after 24 hours and Sutures are removed at clinical control after 14 days and patients are seen again by BCL surgeon after 3 months and are discharged when completely healeddrainage and conventional wound dressing.

INTERVENTIONS:
Device: Prevena™ og ACTIV.A.C™ Therapy System. — A vacuum assisted (negative pressure) system, Prevena ™ and ACTIV.A.C ™ therapy system have been developed to maintain drainage on closed incisions. The system also works by altering the cytokine profile locally so that it functions anti-inflammatory, by increasing local growth factors and promoting angiogenesis19. Negative pressure wound management (NPWM) such as Prevena ™ and ACTIV.AC ™ is a widely used tool with many different variations, but the evidence of effect remains sparse and more studies are required20. We believe that in a dry and closed incision such as the one after BCL surgery, in an area exposed to stretching during healing, it must be an advantage of maintaining drainage, reducing the anti-inflammatory response and increasing angiogenesis.
  Arms: Prevena

SUMMARY:
In a single-blinded randomized, controlled study design the investigators wish to examine to effect of Prevena + ActiV.A.C. therapy system on the postoperative healing in patients operated for chronic pilonidal disease using Bascoms' Cleft Lift procedure. At the department of surgery at The regional Hospital i Randers Denmark the investigators handle cases from the entire region and have a decent patient volume. The investigators have used Bascoms' Cleft left since 2013 and registered complications and experience wound deshisseance or prolonged healing in approx. 15% causing the investigators to challange the postoperative regime.

DETAILED DESCRIPTION:
Background Pilonidal disease (PS) is a common disorder that occurs in the crena ani. A paradigm shift of our perception of the pathology of this disorder has been on its way for several decades and the treatment is slowly starting to follow.

The estimated incidence is 26 per 100,000 although this is subject to large geographical variation. Men present themselves with symptomatic pilonidal disease more than twice as often as women and in population surveys of young students, a 10: 1 male / female ratio has been found, including also asymptomatic pilonidal cysts. The disorder usually affects the younger population with average age at first manifestation of 21 years for men and 19 for women.

Acute manifestations are infected and result in pilonidal abscesses. The treatment of acute abscesses within pilonidal disease is uncontroversial and is based on lateral incision and drainage with subsequent open healing.

The treatment of chronic pilonidal disease, on the other hand, is still controversial. Traditional surgical approach is based on excision of the affected tissue with primary closure or open secondary healing. This treatment, regardless of the manifestation of disease, is characterized by poor healing, complicated postoperative ulceration and recurrence.

Since April 2010, there has been a combination and standardization of the treatment of complicated pilonidal disease at the regional hospital in Randers (Denmark), where patients with 1) recurrence after previous surgery, 2) missing healing > 2 months after surgery and 3) extensive / fistulatory pilonidal disease are offered Bascom's cleft lift (BCL ) operation for the condition.

Bascoms Cleft Lift operation is one of several lateralization techniques that have shown promising results over the last decades. It has the significant advantage compared to the other generally accepted surgical lateralization techniques that it only removed a skin patch (7 mm thick); sub cutis and fat is left in situ regardless of its involvement in the condition: Crena anii is lifted and lateralized, thereby solving the underlying problem and preserving most tissues. The intervention should be significantly less painful than other variants.

In the ongoing work it has been clear that there is delayed healing in a large proportion of these patients by the scheduled postoperative control 14 days after surgery. During the experience of the investigators throughout the first 3 years wound healing complications / delayed healing was found to a variable extent. More than 15% were followed longer than 3 months due to delayed healing and nearly 7% had to be re-operated due to primarily undermining of the cicatrices.

As the operating results are otherwise promising in these recurrent patients, the investigators find it relevant to optimize the postoperative course focusing on better healing.

A vacuum assisted (negative pressure) system, Prevena ™ and ACTIV.A.C ™ therapy system has been developed to maintain drainage on closed incisions. The system also works by altering the cytokine profile locally so that it functions anti-inflammatory, by increasing local growth factors and promoting angiogenesis19. Negative pressure wound management (NPWM) such as Prevena ™ and ACTIV.AC ™ is a widely used tool with many different variations, but the evidence of effect remains sparse and more studies are required. The investigators believe that in a dry and closed incision such as the one after BCL surgery, in an area exposed to stretching during healing, it must be an advantage of maintaining drainage, reducing the anti-inflammatory response and increasing angiogenesis.

Hypothesis

The investigators hypothesize that:

* Patients who have undergone BCL surgery for complicated pilonidal disease have a significantly better healing using Prevena ™ and ACTIV.A.C ™ Therapy System 4-7 days post-operatively compared to patients undergoing normal regimen with drainage and conventional wound dressing.
* That the optimized healing will positively affect the health and wellbeing of patients.

The investigators are not aware of other studies that examine the effect of healing with or without Prevena ™ and ACTIV.A.C ™ or similar devices or its effects on the quality of life of these patients.

Purpose of the study

1. To investigate whether Prevena ™ and ACTIV.A.C ™ Therapy System after BCL surgery for complicated pilonidal disease will improve wound healing compared to a control group of patients treated with conventional drainage and dressing.
2. To examine whether Prevena ™ and ACTIV.A.C ™ treatment and possibly faster healing after surgery for PS affects the self-perceived and pain after surgery using questionnaires / pain journal (Appendix 2 and 3).
3. To describe general health perception among patients with complicated pilonidal disease before and after Bascom's Cleft Lift operation using a questionnaire regarding pilonidal disease.
4. To investigate whether postoperative pain after BCL surgery for complicated pilonidal decreases with Prevena ™ and ACTIV.A.C ™ Therapy System.

Primary end point:

• Evaluate the clinical effect* of Prevena ™ and ACTIV.AC ™ of 4-7 days on BCL cicatrices after 14 days of healing by the following two criteria*: 1) existence of defects in the cicatricees (defects ≤ 5 mm considered fully healed) and 2) undermining of the cicatrices.

Secondary end point:

Evaluate the following short and long term results in connection with BCL surgery and the use of Prevena ™ and ACTIV.A.C ™ Therapy System:

* Symptom related health perception assessed baseline, 14 days postoperatively, after 3 months and after 12 months assessed by questionnaire (Appendix 2)
* Healing after 3 months evaluated according to criteria described above
* Recurrence rate
* Postoperative pain assessed by pain diary (Appendix 3)

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrence after previous surgery for pilonidal disease, cases of poor postoperative healing (> two months) or primary extensive/fistulating disease referred to Randers Regional Hospital for assessment for reconstructive BCL surgery.

Exclusion Criteria:

Patients under 18 years of age

* Patients who smoke (not offered this type of surgery), ceased min. 6 weeks pre-operatively
* Patients with PS lesions are ≤ 3 cm from the anus
* Patients with allergies to Silver or acrylic
* Patients who cannot adhere to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Primary healing | 14 days after surgery
  Evaluation of BCL cicatrices after 14 days of healing by the following two criteria*: 1) existence of defects in the cicatricees (defects ≤ 5 mm considered fully healed) and 2) undermining of the cicatrices.

SECONDARY OUTCOMES:
Health perception | upto 12 months after surgery
  Symptom related health perception assessed baseline, 14 days postoperatively, after 3 months and after 12 months assessed by questionnaire
Long term healing | 3 months after surgery
  Healing after 3 months evaluated according to criteria described previously
early recurrence | up to 12 months after surgery
  record recurrence
post operative pain | 14 days after surgey
  Postoperative pain assessed by pain diary

CONTACTS AND LOCATIONS:
Overall Officials: susanne Haas, Principal Investigator — Clinical officer
Locations (1):
- Regions Hospitalet Randers, Randers, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No
There is not. Data will be handled and analysed within our unit